CLINICAL TRIAL: NCT06051565
Title: Open-label, Single-dose Study of Polysaccharide Superparamagnetic Iron Oxide Injection for Contrast-enhanced Cardiovascular Magnetic Resonance Imaging in Patients With Type 2 Diabetes and Chronic Kidney Disease.
Brief Title: Cardiovascular Contrast-enhanced Magnetic Resonance Imaging Using Polysaccharide Superparamagnetic Iron Oxide Injection in Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DJTCSCYHT-I-03
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2021-10

CONDITIONS: Diabetes; Magnetic Resonance Imaging
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polysaccharide superparamagnetic iron oxide injection (Experimental): Intravenous injected polysaccharide superparamagnetic iron oxide injection at 3 mg/kg dose
  Interventions: Drug: Polysaccharide superparamagnetic iron oxide injection

INTERVENTIONS:
Drug: Polysaccharide superparamagnetic iron oxide injection — Polysaccharide superparamagnetic iron oxide injection can be used for the treatment of iron-deficiency anemia and for magnetic resonance imaging enhancement.

SUMMARY:
This is an open-label, single-center, single-dose study aims to evaluate the effect and safety of polymeric superparamagnetic iron oxide in cardiovascular magnetic resonance imaging for diabetic patients with concomitant chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years, ≤ 80 years.
* Patients who have been diagnosed with chronic kidney disease (CKD) according to diagnostic criteria, meeting at least one CKD diagnostic criterion.
* Patients with a confirmed history of atherosclerosis and/or chronic venous disease (including deep vein thrombosis, thrombotic venous inflammation, lower limb varicose veins, etc.) either in their medical history or diagnosed during hospital admission, and within the past year, at least one imaging examination has confirmed the presence of at least one of the following vascular abnormalities in at least one vascular bed:

  1. ≥50% vascular stenosis;
  2. Arterial aneurysm;
  3. Arterial dissection;
  4. Arteriovenous malformation;
  5. Arteriovenous fistula;
  6. Vascular developmental abnormalities;
  7. Varicose veins, etc. For details, please refer to the inclusion criteria section.
* Patients capable of self-care in daily life.
* Patients who voluntarily agree to participate in this study, sign an informed consent form, have a full understanding of the trial's content, procedures, and potential adverse reactions, and demonstrate good compliance.
* Patients who are unwilling to sign an informed consent form for the exploratory research can still be enrolled in the main study.
* Subjects who have no plans for pregnancy for at least 2 weeks before self-administration of the investigational drug and for at least 6 months after the last use of the investigational drug and voluntarily agree to adopt effective contraceptive measures.

Exclusion Criteria:

* Patients who have undergone stent implantation for vascular treatment in the target vascular bed.
* Patients who have had or currently have malignant tumors within the last 3 years.
* Serum ferritin > 1000 μg/L.
* Patients who are planned to undergo magnetic resonance imaging (MRI) examination for various reasons during the trial.
* Blood donation or significant blood loss (> 450 ml) within the two months before medication.
* Patients with a history of substance abuse involving psychotropic drugs and are unable to quit or have psychiatric disorders.
* Patients with any severe and/or uncontrolled diseases, including:

  1. Outpatients diagnosed through medical history; inpatients diagnosed based on past medical history and current medical history indicating ≥ Grade 2 myocardial ischemia or myocardial infarction, ≥ Grade 2 congestive heart failure (New York Heart Association (NYHA) classification).
  2. Active or uncontrolled severe systemic infections (≥ Common Terminology Criteria for Adverse Events (CTCAE) 5.0 Grade 2).
* Infectious diseases such as cirrhosis, active hepatitis*, syphilis, human immunodeficiency virus (HIV), etc. *Reference for hepatitis B: hepatitis B surface antigen (HBsAg) positive and Hepatitis B Virus (HBV) DNA test value exceeds the upper limit of normal; Reference for hepatitis C: Hepatitis C Virus (HCV) antibody positive and HCV viral titer test value exceeds the upper limit of normal.
* History of immunodeficiency, acquired or congenital immunodeficiency diseases, or organ transplantation.
* Pregnancy or currently breastfeeding or planning to breastfeed during the study.
* Presence of metal objects in the body (dentures, contraceptive rings, metal implants, metal clips, etc.) and claustrophobia.
* Allergic reactions to the investigational drug, its metabolites, or excipients.
* Use of the investigational drug or participation in drug clinical trials within the two months before medication.
* Difficulty with or intolerance to MRI scans.
* Subjects who cannot or will not comply with the hospital management regulations.
* According to the investigator's judgment, patients with accompanying diseases that pose a serious risk to patient safety or may interfere with the completion of the study, or patients deemed unsuitable for inclusion for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The number of vascular segments with lesions | 0 hour after administration
  The number of vascular segments with lesions after administration
Lesion length | 0 hour after administration
  Vascular lesion length
Degree of vascular stenosis | 0 hour after administration
  Vascular stenosis degree

SECONDARY OUTCOMES:
Image quality scores | 0 hour after administration
  Vascular image quality was scored on a 4-point scale. 1 = Vessels not assessable due to poor image quality; 2 = Vessels visualized but only gross features (size/patency) confidently assessable; 3 = Vessels well defined and evaluable for structural pathology with high confidence; 4 = Excellent vessel definition with sharp borders such that fine details can be evaluated with high confidence.
Myocardium T1 values | 0 hour after administration
  Changes from baseline in the longitudinal relaxation value of myocardial tissue.
Signal-to-noise ratio | 0 hour after administration
  The strength of a signal relative to the background noise.
Contrast-to-noise ratio | 0 hour after administration
  The visibility and distinguishability of structures or features of interest in an image in the presence of noise.
Adverse event rate | Baseline up to 24 hours after administration
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Serum iron | Baseline up to 24 hours after administration
  Changes from baseline in the amount of circulating iron that is bound to transferrin and freely circulate in the blood.
Serum ferritin | Baseline up to 30 days and 60 days after administration
  Changes from baseline in the concentration of plasma (or serum) ferritin.
Total iron-binding capacity | Baseline up to 30 days and 60 days after administration
  Changes from baseline in the total amount of iron that can be bound by transferrin proteins in the blood.
Serum transferrin saturation | Baseline up to 30 days and 60 days after administration
  Changes from baseline in the value of serum iron divided by the total iron-binding.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality, China